CLINICAL TRIAL: NCT02720718
Title: Closing the Anastomoses During Laparoscopic Gastric Bypass Surgery: A Comparison of Traditional and Knotless Sutures
Brief Title: Comparison of Laparoscopic Traditional and Knotless Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ St.-Dimpna Geel (Other)
Responsible Party: Principal Investigator, Ben Gys, md, AZ St.-Dimpna Geel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Strat-001
Record Dates: First submitted 2016-03-11; First posted 2016-03-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Anastomosis, Roux-en-Y; Surgical Operation With Anastomosis, Bypass or Graft
Keywords: Gastric Bypass Status for Obesity Complicating Pregnancy, Childbirth and the Puerperium; Laparoscopy; Suture Techniques; Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratafix (Experimental): Patients undergoing laparoscopic RYGB (antecolic, antegastric, "linear anastomosis-technique") using unidirectional barbed (knotless) sutures: Stratafix Unidirectional 2/0.
  Interventions: Device: Stratafix
- Vicryl (Active Comparator): Patients undergoing laparoscopic RYGB (antecolic, antegastric, "linear anastomosis-technique") using classic sutures: Vicryl 2/0.
  Interventions: Device: Vicryl

INTERVENTIONS:
Device: Stratafix
  Arms: Stratafix
Device: Vicryl
  Arms: Vicryl

SUMMARY:
Background

Excess weight and obesity is the fifth leading risk factor for global death. Bariatric surgery is considered as the only effective long-term treatment for morbid obesity. Laparoscopic Roux-en-Y gastric bypass is one of the best surgical procedures, since it achieves excellent long-term results with a low complication rate. Intestinal anastomosis is a very complex and time-consuming procedure in laparoscopy, mainly due to the difficulties of knotting the suture in a limited working area. Barbed sutures may enhance this procedure by eliminating the need for knot tying.

Objective The aim of this study is to compare the safety and efficacy of knotless barbed sutures (Stratafix) and continuous sutures (Vicryl) for closing the gastrojejunal and jejunojejunal anastomosis in obese patients undergoing gastric bypass.

Study design

This is a prospective randomized study. Patients will be randomly assigned to one of two groups: traditional suture group or knotless suture group. Randomization will be realized by sealed envelopes according to a computer-generated sequence of random numbers, which will be opened for the surgeon just before starting the anastomosis. During the surgery the gastrojejunal and jejunojejunal anastomoses will be performed with a stapler (Echelon 45 Endopath) and closed with a traditional (Vicryl) or knotless (Stratafix Unidirectional) suture. The same surgeon, experienced and specialized in laparoscopic gastric bypass technique, will perform all procedures.

Study population

Two hundred patients undergoing laparoscopic Roux-en-Y gastric bypass.

Main study parameters/endpoints

The primary outcome measure will be the rate of anastomosis-related complications (leakage, bleeding, gastric fistula, anastomotic stenosis) at 4 weeks and at 6 months post-op (safety). The secondary outcome measure will be the time spent on closing the gastrojejunal and jejunojejunal anastomosis (efficacy).

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   Obesity

   Excess weight and obesity is the fifth leading risk factor for global death (WHO 2011). It has been demonstrated that conservative treatment of obesity, such as restricting calorie intake, increasing physical activity, and medical treatment, did not succeed in achieving significant long-lasting loss of weight (Flegal 2002). Therefore, bariatric surgery is considered as the only effective long-term treatment for morbid obesity to achieve substantial and sustainable weight loss (Fisher 2002).

   Gastric bypass

   Gastric bypass has a two-way effect: it restricts how much food the stomach can hold (restrictive) and it affects how food and calories are absorbed into the bloodstream (malabsorptive). This combination surgery has the highest success rate for amount of weight loss. Laparoscopic Roux-en-Y gastric bypass is one of the best surgical procedures, since it achieves excellent long-term results with a low complication rate (Schauer 2003, Suter 2011, Fisher 2002). During this procedure two anastomoses - gastrojejunal and jejunojejunal -are constructed. This can be achieved with handsewn suturing or with mechanical stapling (Gonzalez 2003). If the anastomoses are stapled with a linear technique, closing of the enterotomies with sutures is still required. This is a very complex and time-consuming procedure in laparoscopy, mainly due to the difficulties of knotting the suture in a limited working area (De Blasi 2013).

   Knotless sutures

   Barbed sutures may enhance the suturing procedure by eliminating the need for knot tying and by minimizing the help needed from an assistant. However, only a limited number of studies have examined the use of barbed sutures during gastric bypass procedures (De Blasi 2013, Facy 2013, Costantino 2013, Milone 2013). The aim of this study is to compare the safety and efficacy of knotless barbed sutures and traditional continuous sutures for closing the gastrojejunal and jejunojejunal anastomosis after linear stapling in obese patients undergoing gastric bypass.
2. OBJECTIVES

   The aim of this study is to compare the safety and efficacy of knotless barbed sutures (Stratafix Unidirectional) and traditional continuous sutures (Vicryl) for closing the gastrojejunal and jejunojejunal anastomosis in obese patients undergoing gastric bypass.
3. STUDY DESIGN

   This is a prospective randomized study. Patients will be included and enrolled in the study after written informed consent.

   Then, participants will be randomly assigned to one of two groups:
   * Traditional suture group (Vicryl, 2/0)
   * Knotless suture group (Stratafix Unidirectional, 2/0) Randomization will be realized by sealed envelopes according to a computer-generated sequence of random numbers, which will be opened for the surgeon just before starting the anastomosis.

   The surgical procedure will be a standardized laparoscopic Roux-en-Y gastric bypass with the surgeon positioned between the patients legs. During the surgery the gastrojejunal and jejunojejunal anastomoses will be performed with a linear stapler (Echelon 60 EndopathTM) and closed with a traditional (Vicryl) or knotless (Stratafix Unidirectional) suture. The same surgeon, experienced and specialized in laparoscopic gastric bypass technique, will perform all procedures, supported by 1 assistant and 1 research nurse.
4. STUDY POPULATION

   4.1 Population (base) Two hundred patients undergoing a laparoscopic Roux-en-Y gastric bypass at the AZ St. Dimpna in Geel (Belgium).

   4.2 Sample size We have chosen for a sample size of 200 patients (100 in each group). Current literature shows that is a feasible amount of participants for this kind of studies.
5. METHODS

5.1 Study parameters/endpoints

The primary outcome measure will be the rate of anastomosis-related complications (leakage, bleeding, gastric fistula, anastomotic stenosis) for each group:

* At 4 weeks post-op: short-term safety
* At 6 months post-op: long-term safety

The secondary outcome measure will be the time spent on closing the anastomosis (efficacy), measured from first needle in until last knot (Vicryl) or last stitch (Stratafix):

* Gastrojejunal anastomosis
* Jejunojejunal anastomosis

Furthermore, we will register the following co-founders:

* Length of hospital stay
* Total procedure time
* Primary or secondary gastric bypass procedure
* Age
* Gender
* BMI
* ASA score (American Society of Anaesthesiology)
* Co-morbidities (e.g. diabetes)

5.2 Randomisation, blinding and treatment allocation Then, participants will be randomly assigned to one of two groups: traditional suture group or knotless suture group. Randomization will be realized by sealed envelopes according to a computer-generated sequence of random numbers, which will be opened for the surgeon just before starting the anastomosis.

5.3 Study procedures Patients will be included and enrolled in the study after written informed consent.

The surgical procedure will be a standardized laparoscopic Roux-en-Y gastric bypass using a five-port-site technique (2 x 12 mm; 3 x 5 mm), with the following steps:

* Division of the stomach:

  1. Horizontally using a 60-mm regular linear stapler with a blue cartridge (Echelon 60 ENDOPATHTM Stapler Ethicon, Endo-Surgery)
  2. Vertically using two 60-mm regular linear staplers with a blue cartridge (Echelon 60 ENDOPATHTM Stapler Ethicon, Endo-Surgery) to reach the angle of His
* Gastrojejunal anastomosis:

  1. A 60-cm ileal loop is lifted up to the pouch and the anastomosis is performed using 20 mm of a 60-mm regular linear stapler with a blue cartridge (Echelon 60 ENDOPATHTM Stapler Ethicon, Endo-Surgery)
  2. Single-layer continuous suture (Vicryl 2/0 or Stratafix) to close the anastomosis
* Jejunojejunal anastomosis:

  1. The Roux limb is measured at 100 cm (if the patient has a BMI < 50) or at 150 cm (if the patient has a BMI > 50). The anastomosis is performed using a 60-mm regular linear stapler with a white cartridge (Echelon 60 ENDOPATHTM Stapler Ethicon, Endo-Surgery)
  2. Single-layer continuous suture (Vicryl 2/0 or Stratafix) to close the anastomosis
* Completion of bowel division using a 60-mm regular linear stapler with a white cartridge (Echelon 60 ENDOPATHTM Stapler Ethicon, Endo-Surgery)

Afterwards, the mesentery defect and the Petersen's defect are closed using a monofilament non-absorbable suture (Prolene 20). De port sites are not closed.

Patients will be evaluated at 4 weeks and 6 months after the surgery to check for complications.

5.4 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

6. STATISTICAL ANALYSIS

6.1 Descriptive statistics Subject characteristics (age, BMI, co-morbidities) will be described as means ± standard error of the mean for each group. Gender will be described as percentage women for each group.

6.2 Statistical analysis All data will be analyzed using SPSS statistical software.

Continuous variables will be compared amongst the two groups by means of an independent Student's t-test:

* Gastrojejunal anastomosis time
* Jejunojejunal anastomosis time
* Total procedure time
* Length of hospital stay
* Age
* BMI
* ASA score

Categorical variables will be compared by means of a chi-squared test:

* Complication rate
* Primary or secondary gastric bypass
* Gender
* Co-morbidities

A P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* BMI > 40 (morbid obesity) or BMI > 35 with co-morbidities (type 2 diabetes, proven sleep apnoea and/or refractory arterial hypertension)
* Reasonable attempts at other weight loss techniques
* Obesity related health problems
* No psychiatric or drug dependency problems
* Capable to understand the risks and commitment associated with the surgery
* Pregnancy not anticipated in the first two years following surgery

Exclusion Criteria:

* No agreement to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Complication rate. | Up until 6 months after surgery.
  Complications encountered postoperatively: leakage, stenosis, bleeding and gastric fistula.

SECONDARY OUTCOMES:
Length of hospital stay. | Through study completion, an average of 3 days.
  Time between admission and discharge from the hospital.
Total procedure time. | intraoperative
  Time to complete surgery.
Jejunojejunal anastomosis time. | intraoperative
  Time to complete the jejunojejunal anastomosis.
Gastrojejunal anastomosis time. | intraoperative
  Time to complete the gastrojejunal anastomosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Gys, md, Principal Investigator — AZ Sint Dimpna, Geel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costantino F, Dente M, Perrin P, Sarhan FA, Keller P. Barbed unidirectional V-Loc 180 suture in laparoscopic Roux-en-Y gastric bypass: a study comparing unidirectional barbed monofilament and multifilament absorbable suture. Surg Endosc. 2013 Oct;27(10):3846-51. doi: 10.1007/s00464-013-2993-5. Epub 2013 May 31. PMID 23722892
- [Background] De Blasi V, Facy O, Goergen M, Poulain V, De Magistris L, Azagra JS. Barbed versus usual suture for closure of the gastrojejunal anastomosis in laparoscopic gastric bypass: a comparative trial. Obes Surg. 2013 Jan;23(1):60-3. doi: 10.1007/s11695-012-0763-4. PMID 22968833
- [Background] Facy O, De Blasi V, Goergen M, Arru L, De Magistris L, Azagra JS. Laparoscopic gastrointestinal anastomoses using knotless barbed sutures are safe and reproducible: a single-center experience with 201 patients. Surg Endosc. 2013 Oct;27(10):3841-5. doi: 10.1007/s00464-013-2992-6. Epub 2013 May 14. PMID 23670743
- [Background] Fisher BL, Schauer P. Medical and surgical options in the treatment of severe obesity. Am J Surg. 2002 Dec;184(6B):9S-16S. doi: 10.1016/s0002-9610(02)01173-x. PMID 12527344
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Gonzalez R, Lin E, Venkatesh KR, Bowers SP, Smith CD. Gastrojejunostomy during laparoscopic gastric bypass: analysis of 3 techniques. Arch Surg. 2003 Feb;138(2):181-4. doi: 10.1001/archsurg.138.2.181. PMID 12578417
- [Background] Milone M, Di Minno MN, Galloro G, Maietta P, Bianco P, Milone F, Musella M. Safety and efficacy of barbed suture for gastrointestinal suture: a prospective and randomized study on obese patients undergoing gastric bypass. J Laparoendosc Adv Surg Tech A. 2013 Sep;23(9):756-9. doi: 10.1089/lap.2013.0030. Epub 2013 Jul 16. PMID 23859743
- [Background] Schauer PR, Burguera B, Ikramuddin S, Cottam D, Gourash W, Hamad G, Eid GM, Mattar S, Ramanathan R, Barinas-Mitchel E, Rao RH, Kuller L, Kelley D. Effect of laparoscopic Roux-en Y gastric bypass on type 2 diabetes mellitus. Ann Surg. 2003 Oct;238(4):467-84; discussion 84-5. doi: 10.1097/01.sla.0000089851.41115.1b. PMID 14530719
- [Background] Suter M, Donadini A, Romy S, Demartines N, Giusti V. Laparoscopic Roux-en-Y gastric bypass: significant long-term weight loss, improvement of obesity-related comorbidities and quality of life. Ann Surg. 2011 Aug;254(2):267-73. doi: 10.1097/SLA.0b013e3182263b66. PMID 21772127
- [Derived] Gys B, Gys T, Lafullarde T. The Use of Unidirectional Knotless Barbed Suture for Enterotomy Closure in Roux-en-Y Gastric Bypass: a Randomized Comparative Study. Obes Surg. 2017 Aug;27(8):2159-2163. doi: 10.1007/s11695-017-2628-3. PMID 28281235
- See also: World Health Organization. Fact sheet number 311. 2011. — http://www.who.int/mediacentre/factsheets/fs311/en/